CLINICAL TRIAL: NCT04372589
Title: Antithrombotic Therapy to Ameliorate Complications of COVID-19 (ATTACC), in Collaboration With Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV-4)
Brief Title: Antithrombotic Therapy to Ameliorate Complications of COVID-19 (ATTACC)
Acronym: ATTACC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTACC; OZM-113 (Other: Ozmosis Research Inc)
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Pragmatic, Bayesian adaptive randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): Participants randomized to the investigational arm will receive therapeutic anticoagulation for 14 days (or until hospital discharge or liberation from supplemental oxygen >24 hours if previously required, whichever comes first) with heparin, with preference for subcutaneous low molecular weight heparin (enoxaparin preferred, although dalteparin or tinzaparin are also acceptable, as available) if no contraindication is present; alternatively, intravenous unfractionated heparin infusion may be used.
  Interventions: Drug: Heparin
- Control arm (No Intervention): Participants will receive usual care of thromboprophylactic dose anticoagulation according to local practice.

INTERVENTIONS:
Drug: Heparin — Low molecular weight heparin (LMWH) Preferred therapeutic anticoagulant is enoxaparin. Generally regimens: 1.5 mg/kg subcutaneous once daily or 1 mg/kg subcutaneous twice daily. Alternatively, other subcutaneous LMWH used, including tinzaparin (175 anti-Xa IU/kg subcutaneous once daily) or dalteparin (200 IU/kg subcutaneous once daily or 100 IU/kg subcutaneous twice a day).
  Unfractionated heparin (UFH) Commenced, administered, and monitored according to local hospital policy, and guidelines that are used for the treatment of venous thromboembolism (i.e. not for acute coronary syndrome). Intravenous infusion of UFH is according to total body weight and pragmatically adjusted according to local institutional policy to achieve an activated partial thromboplastin time (aPTT) of 1.5-2.5x the reference value. If UFH is used, the availability of a local hospital policy that has specifies an aPTT target in this range or an anti-Xa value is a requirement.
  Arms: Investigational arm

SUMMARY:
Endothelial injury as a consequence of SARS-CoV-2 infection leads to a dysregulated host inflammatory response and activation of coagulation pathways. Macro- and micro-vascular thrombosis may contribute to morbidity, organ failure, and death. Therapeutic anticoagulation with heparin may improve clinical outcomes in patients with COVID-19 through anti-thrombotic, anti-inflammatory, and anti-viral activities of heparins. This pragmatic, Bayesian adaptive randomized controlled trial will determine whether therapeutic anticoagulation with heparin (subcutaneous low molecular weight heparin or intravenous unfractionated heparin) versus usual care reduces the need for intubation or death in hospitalized patients with COVID-19. The trial uses an adaptive design which was chosen to overcome limitations in available data to inform a priori estimation of event rates and possible effect sizes. The adaptive design also includes response-adaptive randomization based on baseline D-dimer level, probing for differential efficacy across subgroups defined based on initial D-dimer level. This Bayesian adaptive randomized trial will stop at a conclusion 1) when the posterior probability that the proportional odds ratio is greater than 1.0 reaches 99% (definition of benefit); 2) when the posterior probability that the proportional odds ratio is greater than 1.2 is less than 10% (definition of futility) or; 3) when the posterior probability that the proportional odds ratio is less than 1.0 is greater than 90% (definition of harm). The trial will enroll a maximum of 3,000 patients, although in many simulations the trial may require fewer patients. The trial is strategically aligned with the international REMAP-CAP/COVID platform trial to accelerate evidence generation.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentre, Bayesian adaptive randomized clinical trial to establish whether therapeutic-dose parenteral anticoagulation improves outcomes for patients hospitalized with COVID-19 (e.g., reduces intubation or mortality). Participants will be randomized either to the investigational arm (therapeutic anticoagulation with heparin for 14 days or until "recovery" [defined as hospital discharge or liberation from supplemental oxygen if initially required], whichever comes first), or to the control arm (usual care, including thromboprophylactic dose anticoagulation according to local practice).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age providing (possibly through a substitute decision maker) informed consent who require hospitalization anticipated to last ≥72 hours, for microbiologically-confirmed COVID-19, enrolled < 72 hours of hospital admission or of COVID-19 confirmation

• If the patient is already hospitalized and the COVID-19 diagnosis is due to an outbreak or an incidental finding, then enrollment can occur within 72 hours of a clinical syndrome attributable to COVID-19 that requires continued hospitalization (e.g. new or worsening oxygen requirements or acute kidney injury) which is further anticipated to extend the hospital admission by an additional 72 hours from randomization.

Exclusion Criteria:

1. Patients admitted to an ICU AND receiving organ support (i.e. high flow nasal oxygen, receiving non-invasive or invasive mechanical ventilation, or are requiring vasopressor/inotrope)
2. Patients for whom the intent is to not use pharmacologic thromboprophylaxis
3. Active bleeding
4. Risk factors for bleeding, including:

   1. intracranial surgery or stroke within 3 months;
   2. history of intracerebral arteriovenous malformation;
   3. cerebral aneurysm or mass lesions of the central nervous system;
   4. intracranial malignancy
   5. history of intracranial bleeding
   6. history of bleeding diatheses (e.g., hemophilia)
   7. history of gastrointestinal bleeding within previous 3 months
   8. thrombolysis within the previous 7 days
   9. presence of an epidural or spinal catheter
   10. recent major surgery <14 days
   11. uncontrolled hypertension (sBP >200 mmHg, dBP >120 mmHg)
   12. other physician-perceived contraindications to anticoagulation
5. Platelet count <50 x10^9/L, INR >2.0, or baseline aPTT >50 (if available per SOC testing)
6. Hemoglobin <80 g/L (to minimize the likelihood of requiring red blood cell transfusion if potential bleeding were to occur)
7. Acute or subacute bacterial endocarditis
8. History of heparin induced thrombocytopenia (HIT) or other heparin allergy including hypersensitivity
9. Current use of dual antiplatelet therapy
10. Patients with an independent indication for therapeutic anticoagulation
11. Patients in whom imminent demise is anticipated and there is no commitment to active ongoing intervention
12. Anticipated transfer to another hospital that is not a study site within 72 hours
13. Enrollment in other trials related to anticoagulation or antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Mortality and days free of organ support | 21 days
  The primary endpoint in the trial is days alive and free of organ support at day 21. This endpoint is defined as the number of days that a patient is alive and free of organ support through the first 21 days after trial entry. Organ support is defined as receipt of invasive or non-invasive mechanical ventilation, high flow nasal oxygen (>30 L/min), vasopressor therapy, or ECMO support. Death at any time (including beyond 21 days) during the index hospital stay is assigned the worst possible score of -1.

SECONDARY OUTCOMES:
Arterial and venous thrombotic conditions | 28 days and 90 days
  A composite endpoint of death, deep vein thrombosis, pulmonary embolism, systemic arterial thromboembolism, myocardial infarction, or ischemic stroke collected during hospitalization or at 28 days and 90 days after enrollment (whichever is earlier).
Intubation and mortality | 30 days
  Ordered categorical endpoint with three possible outcomes based on the worst status of each patient through day 30 following randomization: no invasive mechanical ventilation, invasive mechanical ventilation, or death.
All-cause mortality | 28 days and 90 days
Intubation | 30 days
  Invasive mechanical ventilation.
Hospital-free days | 28 days
  Days alive outside of the hospital through 28 days following randomization.
Ventilator-free days | 28 days
  Days alive not on a ventilator assessed at 28 days following randomization.
Myocardial infarction | 28 days and 90 days
Ischaemic stroke | 28 days and 90 days
Venous thromboembolism | 28 days and 90 days
  Symptomatic proximal venous thromboembolism (DVT or PE).
Vasopressor-free days | 28 days
  Days alive not on a vasopressor assessed at 28 days following randomization.
Renal replacement free days | 28 days
  Days alive not on renal replacement assessed at 28 days following randomization.
Hospital re-admission | 28 days
  Hospital re-admission within 28 days.
Acute kidney injury | Duration of study
  As defined by KDIGO criteria.
Systemic arterial thrombosis or embolism | 28 days and 90 days
ECMO support | Duration of study
  Use of extracorporeal membrane oxygenation (ECMO) support.
Mechanical circuit thrombosis | Duration of study
  Dialysis or ECMO.
WHO ordinal scale | 28 days
  Peak scale over 28 days, scale at 14 days, and proportion with improvement by at least 2 categories compared to enrollment, at 28 days.
Major bleeding | Intervention period (maximum 14 days)
  As defined by the International Society on Thrombosis and Haemostasis (ISTH).
Heparin-induced thrombocytopenia (HIT) | Intervention period (maximum 14 days)
  Laboratory-confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R. Lawler, MD, MPH, Principal Investigator — Peter Munk Cardiac Centre/University Health Network; Ewan C. Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto; Ryan Zarychanski, MD, MSc, Principal Investigator — University of Manitoba
Locations (60):
- United States (13):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic, Jefferson, Louisiana
  - Maine Medical Center, Portland, Maine
  - Henry Ford University, Dearborn, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University School of Medicine/Saint Louis Veterans Affairs Medical Center, St Louis, Missouri
  - Cooper University Health Care, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Montefiore-Einstein Center for Heart and Vascular Care, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Brazil (28):
  - Hospital Unimed do Cariri, Juazeiro do Norte, Ceará
  - Santa Casa de Misericordia de Itabuna, Itabuna, Estado de Bahia
  - Instituto Goiano de Oncologia e Hematologia - INGOH, Goiânia, Goiás
  - Centro de Pesquisas Clínicas Humap - UFMS, Campo Grande, Mato Grosso do Sul
  - Clinica de Campo Grande S/A, Campo Grande, Mato Grosso do Sul
  - Unimed Campo Grande, Campo Grande, Mato Grosso do Sul
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas da UFPR, Curitiba, Paraná
  - Pontifícia Universidade Católica do Paraná, Curitiba, Paraná
  - Parana Medical Research Center, Maringá, Paraná
  - Hospital Agamenon Magalhaes, Recife, Pernanbuco
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Medicina Vascular, Porto Alegre, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Instituto de Cardiologia de Santa Catarina, São José, Santa Catarina
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo, São Paulo
  - Instituto de Molestias Cardio Vasculares de Tatui, Tatuí, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Hospital 9 de Julho, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Instituto de Infectologia Emilio Ribas, São Paulo
  - Instituto do Coração do Estado de São Paulo, São Paulo
  - Sociedade Beneficente Israelita Hospital Albert Einstein, São Paulo
- Canada (16):
  - Victoria General Hospital, Victoria, British Columbia
  - Health Sciences Center Winnipeg, Winnipeg, Manitoba
  - Grace General Hospital, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-University Laval, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (CRIUCPQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
- Mexico (3):
  - Hospital de Infectolog´ñia Centro Médico Nacional La Raza, Azcapotzalco, Mexico City
  - Hospital General Regional 1 Carlos MacGregor Sánchez Navarro, Benito Juárez, Mexico City
  - Hospital General regional 2 El Marqués, Querétaro

REFERENCES:
- [Derived] Wahid L, Froess JD, Ortel TL, Zarychanski R, Berger JS, Cushman M, Angus DC, Renard V, Farahani P, Webb S, Heath A, Godoy LC, Farkouh ME, Hochman JS, Neal MD, Lawler PR. On-Treatment Change in d-Dimer Is Associated With Differential Outcomes Among Therapeutic Dose Heparin-Treated Noncritically Ill Patients Hospitalized for COVID-19. Arterioscler Thromb Vasc Biol. 2025 Jan;45(1):162-164. doi: 10.1161/ATVBAHA.124.321108. Epub 2024 Dec 5. PMID 39633573
- [Derived] Goligher EC, Lawler PR, Jensen TP, Talisa V, Berry LR, Lorenzi E, McVerry BJ, Chang CH, Leifer E, Bradbury C, Berger J, Hunt BJ, Castellucci LA, Kornblith LZ, Gordon AC, McArthur C, Webb S, Hochman J, Neal MD, Zarychanski R, Berry S, Angus DC; REMAP-CAP, ATTACC, and ACTIV-4a Investigators. Heterogeneous Treatment Effects of Therapeutic-Dose Heparin in Patients Hospitalized for COVID-19. JAMA. 2023 Apr 4;329(13):1066-1077. doi: 10.1001/jama.2023.3651. PMID 36942550
- [Derived] REMAP-CAP Investigators; ACTIV-4a Investigators; ATTACC Investigators; Goligher EC, Bradbury CA, McVerry BJ, Lawler PR, Berger JS, Gong MN, Carrier M, Reynolds HR, Kumar A, Turgeon AF, Kornblith LZ, Kahn SR, Marshall JC, Kim KS, Houston BL, Derde LPG, Cushman M, Tritschler T, Angus DC, Godoy LC, McQuilten Z, Kirwan BA, Farkouh ME, Brooks MM, Lewis RJ, Berry LR, Lorenzi E, Gordon AC, Ahuja T, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Contreras A, Costantini TW, de Brouwer S, Detry MA, Duggal A, Dzavik V, Effron MB, Eng HF, Escobedo J, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Froess JD, Fu Z, Galanaud JP, Galen BT, Gandotra S, Girard TD, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Haniffa R, Hegde SM, Hendrickson CM, Higgins AM, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Huang DT, Hudock K, Hunt BJ, Husain M, Hyzy RC, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski A, King AJ, Knudson MM, Kornblith AE, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Gallego Lima F, Linstrum K, Litton E, Lopez-Sendon J, Lother SA, Marten N, Saud Marinez A, Martinez M, Mateos Garcia E, Mavromichalis S, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nicolau JC, Nunez-Garcia B, Park JJ, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Pompilio M, Quigley JG, Rosenson RS, Rost NS, Rowan K, Santos FO, Santos M, Santos MO, Satterwhite L, Saunders CT, Schreiber J, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Singhal AB, Slutsky AS, Solvason D, Stanworth SJ, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Widmer RJ, Wilson JG, Yuriditsky E, Zhong Y, Berry SM, McArthur CJ, Neal MD, Hochman JS, Webb SA, Zarychanski R. Therapeutic Anticoagulation with Heparin in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):777-789. doi: 10.1056/NEJMoa2103417. Epub 2021 Aug 4. PMID 34351722
- [Derived] ATTACC Investigators; ACTIV-4a Investigators; REMAP-CAP Investigators; Lawler PR, Goligher EC, Berger JS, Neal MD, McVerry BJ, Nicolau JC, Gong MN, Carrier M, Rosenson RS, Reynolds HR, Turgeon AF, Escobedo J, Huang DT, Bradbury CA, Houston BL, Kornblith LZ, Kumar A, Kahn SR, Cushman M, McQuilten Z, Slutsky AS, Kim KS, Gordon AC, Kirwan BA, Brooks MM, Higgins AM, Lewis RJ, Lorenzi E, Berry SM, Berry LR, Aday AW, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Costantini TW, de Brouwer S, Derde LPG, Detry MA, Duggal A, Dzavik V, Effron MB, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Galanaud JP, Galen BT, Gandotra S, Garcia-Madrona S, Girard TD, Godoy LC, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Hamburg NM, Haniffa R, Hanna G, Hanna N, Hegde SM, Hendrickson CM, Hite RD, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Hudock K, Hunt BJ, Husain M, Hyzy RC, Iyer VN, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski AL, King AJ, Knudson MM, Kornblith AE, Krishnan V, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Lima FG, Linstrum K, Litton E, Lopez-Sendon J, Lopez-Sendon Moreno JL, Lother SA, Malhotra S, Marcos M, Saud Marinez A, Marshall JC, Marten N, Matthay MA, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Moore SC, Morillo Guerrero R, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nunez-Garcia B, Pandey A, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Perez Gonzalez YS, Pompilio M, Prekker ME, Quigley JG, Rost NS, Rowan K, Santos FO, Santos M, Olombrada Santos M, Satterwhite L, Saunders CT, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Shankar-Hari M, Sheehan JP, Singhal AB, Solvason D, Stanworth SJ, Tritschler T, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Wells BJ, Widmer RJ, Wilson JG, Yuriditsky E, Zampieri FG, Angus DC, McArthur CJ, Webb SA, Farkouh ME, Hochman JS, Zarychanski R. Therapeutic Anticoagulation with Heparin in Noncritically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):790-802. doi: 10.1056/NEJMoa2105911. Epub 2021 Aug 4. PMID 34351721
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- [Derived] Houston BL, Lawler PR, Goligher EC, Farkouh ME, Bradbury C, Carrier M, Dzavik V, Fergusson DA, Fowler RA, Galanaud JP, Gross PL, McDonald EG, Husain M, Kahn SR, Kumar A, Marshall J, Murthy S, Slutsky AS, Turgeon AF, Berry SM, Rosenson RS, Escobedo J, Nicolau JC, Bond L, Kirwan BA, de Brouwer S, Zarychanski R. Anti-Thrombotic Therapy to Ameliorate Complications of COVID-19 (ATTACC): Study design and methodology for an international, adaptive Bayesian randomized controlled trial. Clin Trials. 2020 Oct;17(5):491-500. doi: 10.1177/1740774520943846. Epub 2020 Aug 20. PMID 32815416
- [Derived] Levi M, Thachil J, Iba T, Levy JH. Coagulation abnormalities and thrombosis in patients with COVID-19. Lancet Haematol. 2020 Jun;7(6):e438-e440. doi: 10.1016/S2352-3026(20)30145-9. Epub 2020 May 11. No abstract available. PMID 32407672